CLINICAL TRIAL: NCT01266369
Title: A 12-week With Possible Extension, Prospective, Multicenter, Randomized, Open-label, 2-parallel Group, Phase IIa Study to Compare Efficacy and Safety of AB1010 at 3 or 6 mg/kg/Day in Treatment of Patients With Mastocytosis With Handicap and Bearing Activating Point Mutations in the Phosphotransferase Domain of c-Kit Such as the Main Mutation Asp-816-Val (D816V)
Brief Title: Masitinib in Patients With Mastocytosis With Handicap and Bearing the D816V Mutation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AB Science (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AB06013
Record Dates: First submitted 2010-12-23; First posted 2010-12-24 (Estimated); Last update posted 2018-12-10 (Actual); Status verified 2018-12

CONDITIONS: Mastocytosis
Keywords: mastocytosis; D816V; handicaps
MeSH Terms: conditions — Mastocytosis | interventions — masitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- masitinib 3 mg/kg/day (Experimental): masitinib 3 mg/kg/day
  Interventions: Drug: masitinib
- masitinib 6 mg/kg/day (Experimental): masitinib 6 mg/kg/day
  Interventions: Drug: masitinib

INTERVENTIONS:
Drug: masitinib

SUMMARY:
The objective is to compare efficacy and safety of AB1010 at 3 or 6 mg/kg/day in treatment of patients with mastocytosis with handicap and bearing activating point mutations in the phosphotransferase domain of c-Kit such as the main mutation Asp-816-Val (D816V).

ELIGIBILITY:
Inclusion Criteria:

1. Patients with one of the following documented mastocytosis:

   * Smouldering systemic mastocytosis
   * Indolent systemic mastocytosis with organomegaly
   * Indolent Systemic Mastocytosis having 2 infiltrated organs (skin and bone-marrow)
   * Any mastocytosis with in the last 6 months at least 3 anaphylactic shocks or syncops requiring either use of adrenaline or medical assistance
   * Cutaneous Mastocytosis (CM)
2. Skin biopsy-documented mastocytosis and evaluable disease based upon:

   * Histological criteria: typical infiltrates of mast cells in a multifocal or diffuse pattern in skin biopsy
   * Clinical criteria: typical skin lesions (maculopapular, urticaria pigmentosa, mastocytoma)
3. Missing data (c-kit molecular analysis not done) or documented presence of an activating point mutation in the phosphotransferase domain of c-kit such as D816V c-kit mutation in at least one infiltrated organ (bone marrow or skin)
4. Refractory to at least one of the symptomatic treatments such as:

   * Anti H1
   * Anti H2
   * Proton pump inhibitor
   * Osteoclast inhibitor
   * Cromoglycate Sodium
   * Antileukotriene
   * Other therapies used for the symptomatic care
5. Handicap defined as at least one of the following handicaps:

   * pruritus score ≥ 6
   * number of flushes per week ≥ 7
   * number of stools per day ≥ 4 ,
   * number of mictions per day ≥ 8 ,
   * QLQ-C30 score ≥ 60,
   * Hamilton score ≥ 10

Exclusion Criteria:

1. Patients with one of the following mastocytosis:

   * Systemic Mastocytosis with an Associated clonal Hematologic Non Mast cell lineage Disease (SM-AHNMD)
   * Mast cell leukemia (MCL)
   * Aggressive systemic mastocytosis (ASM)
2. Patient with a major surgery within 2 weeks prior to study entry
3. No vulnerable population will be included in this study

   * Life expectancy < 6 months.
   * Patient is < 5 years free of malignancy, except treated basal cell skin cancer or cervical carcinoma in situ.
   * Patient with grade III/IV cardiac problems as defined by the New York Heart Association Criteria. (i.e., congestive heart failure, myocardial infarction within 6 months of study)
   * Patient has a severe and/or uncontrolled medical disease.
   * Patient has a known diagnosis of human immunodeficiency virus (HIV) infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2007-02; Primary Completion 2007-11 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
efficacy on handicaps | week 12
  Pruritus score at week 12 Number of flushes per week at week 12 Hamilton score at week 12 Fatigue Impact scale at week 12

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Lortholary, MD, PhD, Principal Investigator — Necker Hospital, Paris, France